CLINICAL TRIAL: NCT01525251
Title: The Effect of Nurse Case Manager Model on Caregiver's Adaptation of Disease Uncertainty About Their Child With Neuroblastoma
Brief Title: Nurse Case Manager Model on Neuroblastoma Caregiver's Uncertainty
Acronym: NCMM
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Collaborators: National Science and Technology Council, Taiwan (Other Government); National Taiwan University (Other)
Responsible Party: Principal Investigator, National Taiwan University Hospital, Associate Professor, National Taiwan University Hospital
Other Study IDs: 200907067R
Record Dates: First submitted 2012-01-30; First posted 2012-02-02 (Estimated); Last update posted 2012-02-02 (Estimated); Status verified 2012-01

CONDITIONS: Neuroblastoma
Keywords: primary caregiver; neuroblastoma; support group; posttraumatic stress; uncertainty
MeSH Terms: conditions — Neuroblastoma

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Clinical Problem and Significance: The incidence of neuroblastoma is about 30 cases a year in Taiwan. The five-year survival rate of neuroblastom is near 50% in Taiwan. Compared to the survival rate in Western countries, the treatment in Taiwan needs more efforts to improve. According to the report from the Childhood Cancer Foundation ROC, several children with neuroblastoma did not complete their treatment and or not received the protocol. In addition to the efforts in improving protocol, the reasons for those who drop-out and do not receive complete treatment need the investigators more attention to think of.

Purpose of Study: The main purpose is to evaluate the effects of nurse case manager model on caregivers' adaptation of disease uncertainty about then child with neuroblastorna.

Methods: A longitudinal and prospective design will be used to perform this study. Questionnaire survey and chart review will be the means of data collection for the part of quantative analysis. The qualitative method , semi-structural interview , also will be used to collect data regarding caregiver's perception of social support and adaptation at the same time of self-report of questionnaires survey .There are five points of time to collect data: Baseline (A), 3 months(B) , 6 months(C), 9 months(D),1 year(E) and 1.5 year(F) after eligible subjects agree to participate in the study.

Subjects: The study will use a convenience sample. Once the caregiver's child is on has been diagnosed with neuroblastoma will be recruited in this study.

Instruments: Three Chinese versions of Mishel Uncertainty in Illness-Parent Form , the self-reported socio-demographic questionnaire will be used to collect data. Process recording will be typed once finishing interview for further analysis.

Data Analysis: Quantitative data will be analyzed using SPSS 15.0 statistical software. The data will be analyzed using descriptive statistics and inferred statistics. Content analysis and theme formation will be categorized to assist the interpretation of quantitative results.

Implication: The findings of this study will be expected of the effects of nurse care manager model on children with newoblastoma cancer survivors.

ELIGIBILITY:
Inclusion Criteria:

* Care giver of Neuroblastoma Children

Exclusion Criteria:

* NA

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Caregiver of Neuroblastoma Childern
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2009-08

CONTACTS AND LOCATIONS:
Overall Officials: Ya-Ling Lee, RN,DNSc, Principal Investigator — National Taiwan University
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan, Taiwan